CLINICAL TRIAL: NCT03711318
Title: Buprenorphine Stabilization and Induction Onto Vivitrol for Heroin-dependent Individuals
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: continuing study was no longer feasible
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Alkermes, Inc. (Industry)
Responsible Party: Principal Investigator, Adam Bisaga, Professor of Psychiatry, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7699
Record Dates: First submitted 2018-10-16; First posted 2018-10-18 (Actual); Results first posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-11

CONDITIONS: Heroin Dependence
MeSH Terms: conditions — Heroin Dependence | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Short-term treatment with buprenorphine (Experimental): Short-term treatment with buprenorphine
  Interventions: Drug: Buprenorphine/naloxone

INTERVENTIONS:
Drug: Buprenorphine/naloxone — 3 week treatment with buprenorphine/naloxone

SUMMARY:
A short-term treatment with buprenorphine prior to initiating treatment with naltrexone may increase the proportion of heroin-dependent patients successfully inducted onto Vivitrol.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals between the ages of 18-60
2. Meets DSM-5 criteria of current opioid use disorder with six consecutive months of reported heroin use, supported by a positive urine for opiates indicating regular use of heroin
3. Seeking treatment for opioid use disorder with Vivitrol
4. Capable of giving informed consent and complying with study procedures
5. In otherwise good health based on complete medical history and physical examination, laboratory tests, and EKG
6. BMI between 18-40

Exclusion Criteria:

1. Reported treatment with methadone in the last 3 months or positive urine toxicology for methadone on the day of consent
2. Maintenance on, or regular use of buprenorphine or other prescription opioids
3. Pregnancy, lactation, or failure in a sexually active woman to use adequate contraceptive methods.
4. Active medical illness which might make participation hazardous, such as untreated hypertension, acute hepatitis with AST or ALT > 3 times normal, AIDS (CD4 count under 200 currently or medically ill with an opportunistic infection), unstable diabetes, cardiovascular disease.
5. Active psychiatric disorder which might interfere with participation or make participation hazardous, including DSM-5 Schizophrenia or any psychotic disorder, severe Major Depressive Disorder, or suicide risk or 1 or more suicide attempts within the past year.
6. Physiologically dependent on alcohol or sedative- hypnotics with impending withdrawal. Other substance use diagnoses are not exclusionary.
7. History of allergic or adverse reaction to buprenorphine, naltrexone, naloxone, clonidine, or clonazepam.
8. Chronic neurocognitive disorder
9. History of accidental drug overdose in the last 3 years as defined as an episode of opioid-induced unconsciousness or incapacitation, whether or not medical treatment was sought or received.
10. Painful medical condition that requires ongoing opioid analgesia or anticipated surgery necessitating opioid medications
11. Fentanyl only use, supported by a urine toxicology that is positive for fentanyl only and negative for all other opioids.
12. Court mandated to treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Short-term Treatment With Buprenorphine: Short-term treatment with buprenorphine
  Buprenorphine/naloxone: 3 week treatment with buprenorphine/naloxone followed by initiation of XR-naltrexone
Period: Overall Study
Arm/Group | Short-term Treatment With Buprenorphine
Started | 8
Completed | 1
Not Completed | 7

BASELINE CHARACTERISTICS:
Population: Participants who consented to and initiated study
Arm/Group | Short-term Treatment With Buprenorphine
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 2
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Heroin-dependent Patients Successfully Inducted Onto Vivitrol
Description: Number of patients who received the first Vivitrol injection among those who initiated the induction
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Short-term Treatment With Buprenorphine: Short-term treatment with buprenorphine
  Buprenorphine/naloxone: 3 week treatment with buprenorphine/naloxone followed by initiation of treatment with XR-naltrexone
Arm/Group | Short-term Treatment With Buprenorphine
Number analyzed (Participants) | 8
Participants | 3

ADVERSE EVENTS:
Time Frame: 12 weeks of treatment
Groups:
- Short-term Treatment With Buprenorphine: Short-term treatment with buprenorphine
  Buprenorphine/naloxone: 3 week treatment with buprenorphine/naloxone followed by initiation of treatment with Vivitrol
Arm/Group | Short-term Treatment With Buprenorphine
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Short-term Treatment With Buprenorphine (N=8)
depressive symptoms (Psychiatric disorders) | 1 (1) — patient reported worsening of depressed mood during buprenorphine taper

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/18/NCT03711318/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/18/NCT03711318/SAP_001.pdf